CLINICAL TRIAL: NCT04789486
Title: Nano-SMART: An Adaptive Phase I-II Trial of AGuIX Gadolinium-based Nanoparticles With Stereotactic Magnetic Resonance-guided Adaptive Radiation Therapy for Centrally Located Lung Tumors and Locally Advanced Unresectable Pancreatic Ductal Adenocarcinoma
Brief Title: Nano-SMART: Nanoparticles With MR Guided SBRT in Centrally Located Lung Tumors and Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: NH TherAguix SAS (Other)
Responsible Party: Principal Investigator, Jonathan Leeman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-826
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer; Advanced Pancreatic Adenocarcinoma; Unresectable Pancreatic Cancer; Ductal Adenocarcinoma of the Pancreas
Keywords: Non-small Cell Lung Cancer; Advanced Pancreatic Adenocarcinoma; Unresectable Pancreatic Cancer; Ductal Adenocarcinoma of the Pancreas
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — AGuIX; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- AGUIX + SMART Phase 1 (Experimental): Dose escalation of Activation and Guidance of Irradiation X (AGUIX) and SMART, magnetic resonance imaging (MR)-guided stereotactic body radiation therapy (SBRT).
  Central lung tumor cohort will receive:
  * five fractions of stereotactic body radiation therapy (SBRT)
  * AGuIX Nanoparticle given on -7 or -14 day prior to radiation treatment, then with 1st fraction of radiation and for patients receiving radiation over a two (2) week period with the 4th fraction of radiation .
  Locally advanced/unresectable pancreatic ductal adenocarcinoma-LAPC cohort, will receive:
  five fractions of stereotactic body radiation therapy (SBRT)
  * AGuIX Nanoparticle given on -7 or -14 day prior to radiation treatment, then with 1st fraction of radiation.
  Interventions: Drug: AGuIX; Radiation: Radiotherapy
- AGUIX + SMART Phase 2 (Experimental): Randomized participants will receive recommended phase 1 dose established for their disease group (central lung tumor or locally advanced/unresectable pancreatic ductal adenocarcinoma-LAPC) of Activation and Guidance of Irradiation X (AGUIX) and SMART, magnetic resonance imaging (MR)-guided stereotactic body radiation therapy (SBRT).
  Interventions: Drug: AGuIX; Radiation: Radiotherapy
- SMART Phase 2 (Experimental): Randomized participants will receive standard of care SMART, magnetic resonance imaging (MR)-guided stereotactic body radiation therapy (SBRT).
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Drug: AGuIX — Injected gadolinium-based nanoparticles
  Arms: AGUIX + SMART Phase 1; AGUIX + SMART Phase 2
Radiation: Radiotherapy — Stereotactic magnetic resonance-guided adaptive radiation therapy

SUMMARY:
This research study is being done to help determine the safety and efficacy of gadolinium based nanoparticle, Activation and Guidance of Irradiation X (AGuIX), used in conjunction with MR-guided stereotactic body radiation therapy (SBRT) in the treatment of pancreatic cancer and lung tumors.

DETAILED DESCRIPTION:
This is a seamless phase I/II trial with two separate disease groups/cohorts (centrally located lung tumors and locally advanced/unresectable pancreatic ductal adenocarcinoma-LAPC). The Phase I part is determining for each disease group a safe dose-level that will be evaluated in the Phase II component of the study. The phase II part of the study is a randomized controlled trial that tests, for each disease group, the treatment efficacy of stereotactic body radiation therapy (SBRT) in combination with AGuIX gadolinium-chelated polysiloxane based nanoparticles compared to treatment with stereotactic magnetic resonance (MR)-guided adaptive radiation therapy (SMART) alone

The U.S. Food and Drug Administration (FDA) has not approved Activation and Guidance of Irradiation X (AGuIX) as a treatment for any disease.

AGuIX is a gadolinium-based nanoparticle, gadolinium is the drug used for an MR with contrast. It is believed that the AGuIX may help the radiation received work better by making a tumor more sensitive to the radiation and allowing doctors to see the tumor more clearly. AGuIX has been tested in one previous study with humans. It was found that AGuIX did make tumor cells more sensitive to radiation therapy.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive study treatment for 5 treatment days and will be followed for a year after your treatment ends.

It is expected that about 100 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

Patients should have clinical, radiographical, cytological, or histological confirmation of NSCLC or lung or nodal metastases from another primary cancer defined as within or touching the zone of the proximal bronchial tree, defined as a volume 2 cm in all directions around the trachea and proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus right and left lower lobe bronchi). Tumors that are immediately adjacent (<1 cm) to mediastinal or pericardial pleura or other radiation-sensitive organs such as the esophagus and brachial plexus also are considered central tumors and are eligible for this protocol.

OR Histologically or cytologically confirmed pancreatic ductal adenocarcinoma of the pancreatic head, body or tail.

* Participants must have measurable disease, defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.

Eligible NSCLC patients must have no evidence of nodal involvement (N0), and disease has to be determined unresectable by a thoracic oncologist or the patient is medically inoperable.

* Locally advanced, unresectable pancreatic cancer as determined by a pancreaticobiliary surgeon as part of a multidisciplinary discussion at the investigative site, including multi-phasic CT demonstrating tumor abutment of the SMA or celiac axis, SMV or PV involvement which is not resectable without vascular reconstruction.
* Completion of at least 3 months of standard induction chemotherapy for LAPC, which should consist of either FOLFIRINOX, gemcitabine and nab-paclitaxel, or another standard combination of induction chemotherapy agent, with a washout period no longer than 10 weeks prior to first dose of study drug.
* No evidence of distant metastasis.
* Pancreatic or central NSCLC size ≤ 5cm.
* Age 18 years or older.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Ability to understand and follow the breathing instructions involved in the respiratory gating procedure.
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
* Creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* The effects of AGuIX on the developing human fetus are unknown. For this reason, as well as the known teratogenic effects of radiation, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had prior radiation therapy to the chest or abdomen that would overlap with the current treatment field.
* Participants who are receiving any other investigational agents.
* Participants with known metastatic disease.
* History of allergic reactions attributed to gadolinium-based IV contrast.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because AGuIX is contrast agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AGuIX, breastfeeding should be discontinued if the mother is treated with AGuIX.
* Severe claustrophobia or anxiety.
* Known HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AGuIX. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Active duodenal or gastric ulcer disease or evidence of tumor invasion of the bowel or stomach based on endoscopy.
* Presence of a duodenal stent.
* Unable to undergo magnetic resonance imaging (MRI) due to any of the following:

  1. Presence of MRI-incompatible metal material or devices in the human body
  2. MRI-incompatible Pacemaker or defibrillator
  3. Insulin pump
  4. Aneurysm clip
  5. Artificial heart valve
  6. Cochlear implant
  7. Shrapnel or gunshot injury
  8. Cataract surgery with implant unsafe for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) Phase 1 | 3 months
  Evaluated by the occurrence of Dose Limiting Toxicity (DLT) over the duration of the study using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Compare Local Control at 12 months of Maximum tolerated dose MTD - Phase 2 | 12 months
  Evaluate SMART + AGuIX local control at 12 months compared to SMART alone. Local control at 12 months is defined as the treated tumor is equal to or less than the tumor volume at start of SMART. Progression would be defined per RECIST criteria

SECONDARY OUTCOMES:
Progression-free survival (PFS) at Maximum tolerated dose (MTD) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Assessed by RECIST criteria
Overall Response Rate (ORR) at Maximum tolerated dose (MTD) | Enrollment through study completion, an average of 1 year
  Assessed by RECIST criteria
Serious Adverse Events at 90 Days | 90 days
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used.
Serious Adverse Events at 12 months | 12 months
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used.
Tumor Changes | Enrollment through study completion, an average of 1 year
  Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
Compare disease-specific survival | Enrollment through study completion, an average of 1 year
  Bayesian hierarchical two-sample test for binary outcomes
compare R0 resection rate | Enrollment through study completion, an average of 1 year
  Bayesian hierarchical two-sample test for binary outcomes
Compare overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Bayesian hierarchical two-sample test for binary outcomes
Quality of Life (QoL)-Performance Status utilizing PROMIS Physical and Mental Health batteries | Baseline through study completion, an average of 1 year
  Described using descriptive statistics and longitudinal analyses
Quality of Life (QoL)-Completion of Daily Activities utilizing PROMIS Physical and Mental Health batteries | Baseline through study completion, an average of 1 year
  Described using descriptive statistics and longitudinal analyses

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leeman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu